CLINICAL TRIAL: NCT04033250
Title: Personalized Colonoscopy Preparation for Patients With Risk Factors for Inadequate Preparation: A Randomized Control Trial
Brief Title: Personalized Colonoscopy Preparation for Patients With Risk Factors for Inadequate Preparation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Amir Klein MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0117-19-RMB CTIL
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Inadequate Preparation for Colonoscopy; Personalized Colonoscopy Preparation
MeSH Terms: interventions — picosulfate sodium; Magnesium Oxide; Citric Acid; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional arm (group A) (Experimental): Patients with risk factors for IBP who will receive "intensified" bowel preparation
  Interventions: Drug: Sodium Picosulfate / Magnesium Oxide / Citric Acid in two split doses + one dose of polyethylene glycol + two Bisacodyl tablets day before the procedure
- Control arm (group B) (Active Comparator): Patients with risk factors for IBP who will receive standard bowel preparation
  Interventions: Drug: Sodium Picosulfate / Magnesium Oxide / Citric Acid in two split doses + one dose of polyethylene glycol + two Bisacodyl tablets day before the procedure
- Control arm (group c) (Active Comparator): Patients without risk factors for IPB who will receive standard bowel preparation
  Interventions: Drug: Sodium Picosulfate / Magnesium Oxide / Citric Acid in two split doses + one dose of polyethylene glycol + two Bisacodyl tablets day before the procedure

INTERVENTIONS:
Drug: Sodium Picosulfate / Magnesium Oxide / Citric Acid in two split doses + one dose of polyethylene glycol + two Bisacodyl tablets day before the procedure — Bowel preparation
  Other Names: Sodium Picosulfate / Magnesium Oxide / Citric Acid in two split doses

SUMMARY:
Adequate bowel preparation is one of the most important quality measures in colonoscopy. Previous studies identified several factors associated with inadequate bowel preparation (IBP). No study has attempted to assign a different regimen to patients based on the presence of risk factors for inadequate bowel preparation.

The aim of the study is to check if a personalized bowel preparation regimen based on risk factors for IBP, will lead to an overall improvement in bowel preparation during colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* previous IBP
* concurrent medical conditions (e.g. diabetes, constipation)
* medications (e.g. opioids and tricyclic antidepressants)

Exclusion Criteria:

* previous colonic resection
* patients with IBD
* active CRC
* chronic kidney disease at any stage
* congestive heart failure at any stage
* liver cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Improved bowel preparation | Index colonoscopy
  Boston Bowel Preparation Scale at index colonoscopy will be measured. The grading is between 1 and 3 for each segment of colon (ascending, transverse, descending) where 1 is poor and 3 is excellent (subscale). The final score is between 3 and 9 summing up the scores for each segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam MC, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No